CLINICAL TRIAL: NCT01981668
Title: The JET Study: a Phase I Trial of Cabazitaxel, Radiotherapy and Long-term Androgen Deprivation
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: no Canadian centre interested in conducting study in a reasonable timeframe
Sponsor: Nova Scotia Cancer Centre (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Derek R Wilke MD,MSc,FRCPC, Research Director, Nova Scotia Cancer Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CABAZ-L-06233
Record Dates: First submitted 2013-10-29; First posted 2013-11-11 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cabazitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cabazitaxel, Eligard and Radiotherapy (Experimental): This study utilizes a conventional phase I study design with a '3+3 cohort expansion' design(15), to determine the MTD of 1) Cabazitaxel, in Part A, and 2) Radiotherapy, in Part B. The determination of the MTD is given in Section 5.2, Definition of Dose - Limiting Toxicity. All patients who enter the study, and begin concurrent chemo-radiation are analyzable for the primary endpoint of the study.
  Interventions: Drug: cabazitaxel

INTERVENTIONS:
Drug: cabazitaxel — Concurrent cabazitaxel, radiotherapy and Eligard for 3 years
  Other Names: Jevtana

SUMMARY:
This study utilizes a conventional phase I study design with a '3+3 cohort expansion' design(15), to determine the maximum tolerated dose(MTD) of 1) Cabazitaxel, in Part A, and 2) Radiotherapy, in Part B. The determination of the MTD is given in Section 5.2, Definition of Dose - Limiting Toxicity. All patients who enter the study, and begin concurrent chemo-radiation are analyzable for the primary endpoint of the study.

DETAILED DESCRIPTION:
This study utilizes a conventional phase I study design with a '3+3 cohort expansion' design(15), to determine the maximum tolerated dose(MTD) of 1) Cabazitaxel, in Part A, and 2) Radiotherapy, in Part B. The determination of the MTD is given in Section 5.2, Definition of Dose - Limiting Toxicity. All patients who enter the study, and begin concurrent chemo-radiation are analyzable for the primary endpoint of the study.

Assuming that dose-limiting toxicity is not encountered, and both the maximum dose of Cabazitaxel is reached, in Part A of the study, and the maximum dose of Radiotherapy is reached in Part B of the study, the maximum number of patients required is as follows: Clinical Study Protocol - The JET study Date: September 11, 2012 Part A: 3 patients per level x 5 levels, plus 3 patients (for a total of 6) at the highest dose level of Cabazitaxel = 15 + 3 = 18 Part B: 3 patients per level x 3 levels, plus 3 patients (for a total of 6) at the highest dose level of Radiotherapy = 9 + 3 = 12 The total number of patients required is 30. Patients that do not complete concurrent chemotherapy, radiotherapy, and androgen deprivation therapy, for reasons other than DLT will be replaced.

Given our experience in chemo-radiation studies in a similar patient population, our Centre is anticipated to accrue 3 patients per month.

ELIGIBILITY:
Inclusion Criteria:

* High risk prostate cancer

Exclusion Criteria:

* mets

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Toxicity | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Derek R Wilke, MD,MSc,FRCPC, Principal Investigator — department of radiation oncology